CLINICAL TRIAL: NCT03665909
Title: A Proactive Health Monitoring Intervention for Dementia Caregivers: The eNeighbor
Brief Title: A Proactive Health Monitoring Intervention for Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1401547541; R18HS022836 (AHRQ)
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote activity monitoring (Experimental): Receive the remote activity monitoring system (i.e., "eNeighbor;" see intervention description) over an 18-month period.
  Interventions: Other: Remote activity monitoring system
- Control (No Intervention): Control participants do not receive the remote activity monitoring intervention.

INTERVENTIONS:
Other: Remote activity monitoring system — The home-based sensor technology of eNeighbor relies on multiple, non-invasive and safe remote monitors (up to 6 sensors) that can alert family caregivers and/or health professionals to potentially negative situations that lead to adverse outcomes (e.g., wandering, falls, incomplete activity of daily living tasks). The technology platform of eNeighbor relies on wireless infrastructure that allows for remote monitoring via alerts that are communicated to the family caregiver's or nurse care manager's personal computers or handheld devices. The Alerts that are generated from the sensors detected abnormal motion or activity are sent to the family caregiver as well as a nurse care manager that monitors the real-time information generated by the eNeighbor sensors.
  Other Names: eNeighbor
  Arms: Remote activity monitoring

SUMMARY:
The objective of this 5-year demonstration project is to build on the work of The Lutheran Home Association (TLHA) and conduct an embedded experimental mixed methods evaluation to determine the efficacy of the eNeighbor technology in improving outcomes among persons with Alzheimer's disease or related dementias (ADRD) living in the community and their family caregivers. The Specific Aims are as follows: 1) To compare 100 ADRD caregivers randomly assigned to an attention control with 100 ADRD caregivers who utilize eNeighbor over an 18-month period to determine if the use of the remote sensor technology results in a) significant (p < .05) increases in caregiver self-efficacy and sense of competence, b) significant decreases in caregiver distress (subjective stress, depressive symptoms), c) significant delays of or reductions in negative health transitions (falls, wandering events) and service utilization (residential care placement, hospitalizations) for persons with ADRD; and d) greater cost-effectiveness; 2) To determine through "embedded" qualitative data collection components how eNeighbor is successfully utilized and why this health monitoring technology benefits persons with ADRD and their family caregivers; and 3) To engage stakeholders on a quarterly basis throughout this 5-year demonstration project in order to enhance the utility and stakeholder-relevance of health monitoring technology for families who care for persons with ADRD. The investigators anticipate that the successful completion of the project aims will position the eNeighbor as an innovative, stakeholder-centric service that offers robust support for family caregivers of persons with ADRD in the community.

DETAILED DESCRIPTION:
In collaboration with a 15-member Community Advisory Board that includes community care providers, healthcare organizations, and ADRD caregivers themselves, the proposed 5-year project will build on the current efforts of The Lutheran Home Association (TLHA) to evaluate eNeighbor remote monitoring technology for persons with ADRD living in the community and their family caregivers. The Specific Aims are as follows:

1. To determine the efficacy of remote sensor technology over an 18-month period for 100 persons with ADRD and their caregivers randomly assigned to an eNeighbor treatment condition when compared to 100 usual care controls. The investigators hypothesize:

   Hx. 1) Significant (p < .05) improvements in caregiver self-efficacy and sense of competence in managing a relative's ADRD; Hx. 2) Significant reductions in caregiver distress (e.g., subjective stress, or feelings of emotional fatigue and role entrapment; depressive symptoms); Hx. 3) Significant delay of or reductions in health transitions (falls, wandering) and service utilization (hospitalizations, nursing home admission) for persons with ADRD; and Hx. 4) Greater cost-effectiveness associated with a person with ADRD's health service use.
2. To "embed" evaluation components: a) during the randomized controlled evaluation through the administration of open-ended survey items to all ADRD caregivers in the eNeighbor treatment condition every 6 months to examine the utility of the remote health monitoring technology; and b) at the conclusion of the 18-month evaluation by purposively sampling 15 ADRD caregivers who reported positive acceptance on the embedded qualitative and quantitative 6-, 12-, and 18-month system reviews and 15 ADRD caregivers who reported low acceptance on the embedded qualitative and quantitative 6-, 12-, and 18-month system reviews to participate in semi-structured interviews. The interviews will help the research team determine why the health monitoring intervention was or was not efficacious; and
3. To engage stakeholders on a quarterly basis throughout the 5-year project with the goal of enhancing the utility (via community-based participatory approaches) and stakeholder-relevance of eNeighbor implementation and evaluation for family caregivers of persons with ADRD.

ELIGIBILITY:
INCLUSION

* The person with ADRD must be English speaking;
* The person with ADRD must have a physician diagnosis of ADRD (Alzheimer's disease, Lewy Body disease, fronto-temporal dementia, or stroke/vascular dementia; mild cognitive impairment only)
* The person with ADRD must not be currently receiving care or case management services;
* The person with ADRD must be 55 years of age and over;
* The caregiver of persons with ADRD must be English speaking;
* The caregiver of persons with ADRD must be 21 years of age and over;
* The caregiver of persons with ADRD must self-identify as someone who provides help to the person with ADRD because of their cognitive impairments;
* The caregiver of persons with ADRD must self-identify as the person most responsible for providing hands-on care to the person with ADRD;
* The caregiver of persons with ADRD must plan to remain in the area for at least 18 months in order to reduce possible loss to follow-up; and
* The caregiver of persons with ADRD must indicate a willingness to use eNeighbor.

EXCLUSION

● Those who do not meet the above inclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Nursing home utilization at 18 months for the person with ADRD | 18-months
  Caregiver report of nursing home use at 18 months.

SECONDARY OUTCOMES:
Perceptions of change in caregiver self-efficacy | Baseline, 6-months, 12-months, 18-months
  An 8-item survey measure of caregiver self-efficacy. Item responses range from 1 "very unconfident" to 5 "very confident." Scores are summed and can range from a score of 1 (low self-efficacy) to 40 (high self-efficacy).
Perceptions of change in caregiver competence | Baseline, 6-months, 12-months, 18-months
  The 7-item Short Sense of Competence Questionnaire (SSCQ), which assesses individuals' sense of capability in providing assistance to a relative with Alzheimer's disease or related dementias via survey report. Item responses range from 1 = strongly disagree to 5 = strongly agree. Item responses are summed, with a total score range of 5 to 35.
Perceptions of change in caregiver burden | Baseline, 6-months, 12-months, 18-months
  The 22-item Zarit Burden Interview self-report survey measure. Item responses range from 0 "never" to 4 "nearly always." Scores are summed and can range from a score of 0 (no burden) to 88 (high burden).
Perceptions of change in caregiver role captivity | Baseline, 6-months, 12-months, 18-months
  The 4-item role captivity measure assesses the involuntary aspects of the caregiving role. Item responses range from 1 = "not at all" to 4 = "very much." The total role captivity score is the sum of item responses with a range of 4 (no role captivity) to 16 (high role captivity).
Change in caregiver role overload | Baseline, 6-months, 12-months, 18-months
  The 3-item role overload survey measure ascertains caregivers' feelings of emotional and physical fatigue. Item responses range from 1 = "not at all" to 4 = "very much." The total role overload score is the sum iof item responses with a range of 4 (no role overload) to 16 (high role overload).
Change in frequency/perceptions caregiver depressive symptom severity | Baseline, 6-months, 12-months, 18-months
  The 20-item Center for Epidemiological Studies Depression (CES-D) survey measure is used to assess caregivers' depressive symptoms. Item responses range from 1 = "Rarely or none of the time (less than 1 day)" to 5 = "Most of the time (5-7 days)." The total CES-D score is summed, with a range of 20 (little to no depressive symptoms) to 100 (frequent depressive symptoms).
Perceived acceptability/utility of remote activity monitoring at 6-, 12-, and 18-months | 6-months, 12-months, 18-months
  The Remote Activity Monitoring Review Checklist is administered to caregiving participants in the treatment condition at the 6-month, 12-month and 18-month follow-up survey intervals. The checklist consists of 21 self-report survey Likert scale items. Item responses range from 1 = strongly disagree to 5 = strongly agree. The total checklist score is averaged, with a score of 1 = the remote activity monitoring system was not well-received/accepted to 5 = the remote activity monitoring system was very well received/accepted.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell LL, Peterson CM, Rud SR, Jutkowitz E, Sarkinen A, Trost S, Porta CM, Finlay JM, Gaugler JE. "It's Like a Cyber-Security Blanket": The Utility of Remote Activity Monitoring in Family Dementia Care. J Appl Gerontol. 2020 Jan;39(1):86-98. doi: 10.1177/0733464818760238. Epub 2018 Mar 4. PMID 29504488
- [Background] Zmora R, Mitchell LL, Bustamante G, Finlay J, Nkimbeng M, Gaugler JE. Dementia Caregivers' Experiences and Reactions to Remote Activity Monitoring System Alerts. J Gerontol Nurs. 2021 Jan 1;47(1):13-20. doi: 10.3928/00989134-20201208-03. PMID 33377980
- [Result] Gaugler JE, Zmora R, Mitchell LL, Finlay JM, Peterson CM, McCarron H, Jutkowitz E. Six-Month Effectiveness of Remote Activity Monitoring for Persons Living With Dementia and Their Family Caregivers: An Experimental Mixed Methods Study. Gerontologist. 2019 Jan 9;59(1):78-89. doi: 10.1093/geront/gny078. PMID 29982413
- [Result] Gaugler JE, Zmora R, Mitchell LL, Finlay J, Rosebush CE, Nkimbeng M, Baker ZG, Albers EA, Peterson CM. Remote activity monitoring for family caregivers of persons living with dementia: a mixed methods, randomized controlled evaluation. BMC Geriatr. 2021 Dec 18;21(1):715. doi: 10.1186/s12877-021-02634-8. PMID 34922475

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03665909/Prot_SAP_003.pdf